CLINICAL TRIAL: NCT06437951
Title: A Randomized, Double-blind, Placebo-controlled, Single/Multiple-dose, Phase 1 Clinical Trial to Evaluate the Safety/Tolerability and Pharmacokinetics, and Pharmacodynamics After Intravenous DWP14012 Injection in Healthy Participants
Brief Title: to Evaluate the Safety/Tolerability and Pharmacokinetics, and Pharmacodynamics of DWP14012 Injection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWJ1521104
Record Dates: First submitted 2024-05-13; First posted 2024-05-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Erosive Gastroesophageal Reflux Disease
MeSH Terms: interventions — fexuprazan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part1_test group (Experimental): IV injection of test drugs by dose group
  Interventions: Drug: Fexuprazan Injection
- Part1_placebo group (Placebo Comparator): IV injection of test drugs by dose group
  Interventions: Drug: Fexuprazan Injection placebo
- Part2 (Experimental): All Participants take IV injection of test drugs
  Interventions: Drug: Fexuprazan Injection_part 2
- Part3_test group (Experimental): In the case of test group, take IV injection in the period 1 and take a tablet in the period 2
  Interventions: Drug: Fexuprazan Injection_part 3; Drug: Fexuprazan tablet
- Part3_reference group (Active Comparator): In the case of reference group, take a tablet in the period 1 and take IV injection in the period 2
  Interventions: Drug: Fexuprazan Injection_part 3; Drug: Fexuprazan tablet

INTERVENTIONS:
Drug: Fexuprazan Injection — 20/40/80 mg
  Arms: Part1_test group
Drug: Fexuprazan Injection placebo — 20/40/80 mg
  Arms: Part1_placebo group
Drug: Fexuprazan Injection_part 2 — 20mg
  Arms: Part2
Drug: Fexuprazan Injection_part 3 — 40mg
  Arms: Part3_reference group; Part3_test group
Drug: Fexuprazan tablet — 40mg
  Arms: Part3_reference group; Part3_test group

SUMMARY:
to evaluate the safety/tolerability and pharmacokinetics, and pharmacodynamics after intravenous DWP14012 injection in healthy participants

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 19 to 50 at the time of screening tests
2. Those who weigh more than 50.0 kg, 90.0 kg or less, and have a BMI of 18.5 or more and 29.9 or less at the time of screening inspection BMI (kg/m2) = Weight (kg) / {Height (m)}2
3. In the case of female volunteers, those who are not necessarily pregnant or lactating or who are in surgical infertility (bilateral ovarian obstruction, hysterectomy, bilateral ovarian resection, etc.)
4. A person who voluntarily decides to participate after hearing and fully understanding the detailed explanation of this clinical trial and agrees in writing before a screening procedure
5. A person who is suitable for this test when judging the tester by physical examination, clinical laboratory examination, questionnaire, etc

Exclusion Criteria:

1. Clinically significant hepatomegaly (severe liver disorder, viral hepatitis, etc.), kidney (severe renal disorder, etc.), nervous system, immune system, respiratory system, digestive system, endocrine system, blood and tumor, cardiovascular system (heart failure, Torsades de points, etc.), urinary system, mental system (fever disorder, obsessive compulsive disorder, etc.), sexual dysfunction, etc
2. A person who has a history of gastrointestinal diseases (such as Crohn's disease, ulcers, gastritis, gastritis, gastroesophageal reflux disease, etc.) or surgery (except simple appendectomy or hernia) that may affect the safety, pharmacokinetics and pharmacodynamic evaluation of clinical medicines
3. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
4. A person who has been tested positive for Helicobacter pylori
5. Those who have anatomical impairments in insertion and maintenance of the pH meter catheter etc

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
PK of Fexuprazan | 0 and 72hour
  1. Blood and urinary concentrations of Fexuprazan by part
PK of metabolite | 0 and 72hour
  1. Blood and urinary concentrations of metabolite by part
PD of Fexuprazan | up to 15days
  pH monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Injin zhang, Ph.D, Principal Investigator — Seoul National University College of Medicine and Hospital